CLINICAL TRIAL: NCT02427516
Title: Cost of Monitoring Patients Treated With Vitamin K Antagonists in Spain
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Badalona Serveis Assistencials (Other); IMS Health (Other)
Responsible Party: Sponsor
Other Study IDs: CV185-374
Record Dates: First submitted 2015-04-23; First posted 2015-04-28 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Anticoagulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- NVAF-VKA cohort: NVAF patients who initiate a VKA treatment
- VTE-VKA cohort: VTE patients who initiate a VKA treatment

SUMMARY:
To estimate annualized total cost rates (i.e. direct medical costs from hospitalizations, consultations, medications, and tests) of adequately controlling a patient (i.e. INR between 2-3 and TTR≥ 60%) diagnosed with non-valvular atrial fibrillation (NVAF) or venous thromboembolism (VTE), and treated with vitamin K antagonists (VKA) in Spain.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Patients aged 18 or older over the study period
* Patients with a diagnosis for NVAF or VTE anytime in their medical records
* Patients having at least one year of enrolment in the database prior to the index date
* Patients newly initiated with VKA during the study period (index date)

Exclusion Criteria:

* Patients with a diagnosis for both NVAF and VTE anytime in their medical records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with NVAF or VTE and treated with VKA
Sampling Method: Probability Sample
Enrollment: 1144 (Actual)
Dates: Start 2009-01; Primary Completion 2015-05 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Annualized total and per patient cost of patients diagnosed with NVAF or VTE treated with VKA and according to coagulation control status based on electronic clinical records | Approximately 60 months
  Per patient cost: direct medical costs from hospitalizations, consultations, medications, and tests; Coagulation control status: adequately controlled patients defined by INR between 2-3 and TTR≥ 60%

SECONDARY OUTCOMES:
Demographic and clinical characteristics for all patients diagnosed with NVAF or VTE treated with VKA and according to coagulation control status based on electronic clinical records | Approximately 60 months
  Variables measured: age, gender, employment status, smoking status, BMI, major co-morbidities (including CHARLSON index), CHA2DS2-VASc score, presence and frequency of INR measurement, and INR therapeutic range.
Healthcare resource rates for all patients diagnosed with NVAF or VTE treated with VKA and according to coagulation control status based on electronic clinical records | Approximately 60 months
  Healthcare resources used (i.e. hospitalizations, consultations, medication, and tests) by patients will be measured according to coagulation control status. For each healthcare resource the number and percentage of patients using it and the mean, SD, median min, max and valid n will be reported; as well as the number of times that each patient uses the resource.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx